CLINICAL TRIAL: NCT01246011
Title: Significance of Antibodies to Heparin/Platelet Factor 4 Complex in Vein Graft Patency and Potential Role of Argatroban for Prevention of Vein Graft Occlusion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was too slow.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2010P001386
Record Dates: First submitted 2010-11-17; First posted 2010-11-23 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Bypass Graft Surgery; Presence of Heparin/Platelet Factor 4 Antibody
MeSH Terms: interventions — argatroban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Heparin PF4 antibody positive -Drug (argatroban and warfarin) (Experimental): Post-CABG heparin PF4 antibody positive with no signs or symptoms of HIT randomized to receive argatroban and warfarin
  Interventions: Drug: Argatroban and warfarin
- Heparin PF4 antibody positive no drug (No Intervention): Post-CABG heparin PF4 antibody positive with no signs or symptoms of HIT randomized to receive no medication
- Heparin PF4 antibody negative (No Intervention): Post-CABG heparin PF4 antibody negative with no signs or symptoms of HIT randomized to receive no medication

INTERVENTIONS:
Drug: Argatroban and warfarin — Subjects with the presence of heparin PF4 antibodies without signs or symptoms of HIT post CABG will be randomized to receive argatroban and warfarin or no drug for one month.
  Arms: Heparin PF4 antibody positive -Drug (argatroban and warfarin)

SUMMARY:
Heparin/Platelet Factor 4 (PF4) antibody testing will be performed in subjects who have just undergone coronary artery bypass grafting (CABG) surgery. 30 subjects with a positive antibody result and no signs or symptoms of Heparin Induced Thrombocytopenia (HIT) will be randomized to receive argatroban and warfarin. 30 subjects with a positive antibody result and no signs or symptoms of HIT will be randomized to receive no treatment. 30 subjects with a negative antibody result will also be followed in the study. All subjects will have a cardiac CT scan at about 30 days post surgery to measure the patency of their coronary artery bypass vein grafts. This study will evaluate if treating patients who have heparin PF4 antibodies post-CABG with argatroban and warfarin has any effect on the short-term patency of coronary artery bypass vein grafts.

DETAILED DESCRIPTION:
This is a prospective, randomized, single center study. Patients scheduled for CABG will be screened and enrolled. Subjects positive for heparin/PF4 antibody within 24 h after CABG and without clinical suspicion of HIT will be randomized into one of two groups. An additional 30 patients with negative antibody titers will serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for CABG (males or non-pregnant females)
2. > 18 years old with at least one vein graft planned
3. Able to provide written informed consent

Exclusion Criteria:

1. Patients who, in the investigator's or attending surgeon's opinion, are unsuitable for anticoagulation due to their clinical status
2. Documented history of allergy to iodinated contrast media, warfarin, or argatroban
3. Chronic renal impairment with CrCl<60 ml/min
4. Recent bleeding episode
5. Congestive Heart Failure (EF< 30%)
6. Bleeding diathesis or known thrombophilic disorder
7. Atrial fibrillation or other condition requiring anticoagulation at the time of enrollment
8. Documented history of heparin induced thrombocytopenia
9. Clinical suspicion of HIT at the time of randomization, defined as 50% decrease in Platelet count from last heparin exposure or Platelet count <100,000/ml
10. Hepatic dysfunction (defined as LFTs > 3 times the upper limit of normal)
11. Patients with a history of bleeding complications post-CABG
12. Hemorrhagic stroke
13. Gastrointestinal bleeding
14. Requirement for fresh frozen plasma
15. Recent central nervous system or ophthalmic surgery
16. Aneurysm
17. History of psychosis or senility
18. Malignant hypertension
19. Clinically significant pericarditis or pericardial effusion
20. Bacterial endocarditis
21. Hematocrit < 24%
22. Valve replacement or repair at time of CABG
23. Subjects with signs or symptoms of possible Transient Ischemic Attack or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began enrolling in January 2011 and screening ended in July 2011, after it was decided that enrollment was too slow and that the study should be terminated.
Period: Overall Study
Arm/Group | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) | Heparin PF4 Antibody Positive no Drug | Heparin PF4 Antibody Negative
Started | 0 | 0 | 9
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 4
Not completed — If needed warfarin clinically, withdrawn | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) | Heparin PF4 Antibody Positive no Drug | Heparin PF4 Antibody Negative | Total
Number analyzed (Participants) | 0 | 0 | 9 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 5 | 5
  >=65 years |  |  | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 61.9 (11.3) | 61.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 1 | 1
  Male |  |  | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States |  |  | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Coronary Artery Bypass Vein Graft Patency
Description: Vein graft patency as measured by computed tomography
Time Frame: Approximately 30 Days post CABG
Population: No analysis will be done due to early study termination
Arm/Group | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) | Heparin PF4 Antibody Positive no Drug | Heparin PF4 Antibody Negative
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Major Bleeding Events.
Description: Intracranial bleed or any clinically overt sign of hemorrhage that is associated with a fall in hemoglobin > 5 g/dL.
Time Frame: At 2weeks post CABG
Population: No analysis will be done due to early study termination.
Arm/Group | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) | Heparin PF4 Antibody Positive no Drug | Heparin PF4 Antibody Negative
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: 1 subject withdrew from the study prior to having a specimen drawn, so there were only 8 participants at risk
Arm/Group | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) | Heparin PF4 Antibody Positive no Drug | Heparin PF4 Antibody Negative
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 5/8
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) (N=0) | Heparin PF4 Antibody Positive no Drug (N=0) | Heparin PF4 Antibody Negative (N=8)
Hypotension after Coronary Artery Bypass Graft Surgery (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Atrial Fibrillation after Coronary Artery Bypass Surgery (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Bleeding during or immediately after Coronary Artery Bypass Surgery (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heparin PF4 Antibody Positive -Drug (Argatroban and Warfarin) (N=0) | Heparin PF4 Antibody Positive no Drug (N=0) | Heparin PF4 Antibody Negative (N=8)
Low Hematocrit after Coronary Artery Bypass Graft Surgery (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Urinary Retention after Coronary Artery Bypass Surgery (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Post operative nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Back spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Parkinson's-like features (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was ended early due to slow enrollment and results will not be analyzed. The 4 subjects who completed the study were all in the same arm of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes